CLINICAL TRIAL: NCT06113172
Title: Behavior of the Iliofemoral Segment
Acronym: BEHAVIOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 651
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Artery Stenosis
Keywords: iliofemoral segment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Patients referred for endovascular procedure (aortic or peripheral), with an indication of CTA comprising the CFA region, without significant lesions of the external iliac and common femoral arteries. In case of difference of calcifications between both CFA, the CFA with less calcifications will be chosen for analysis.
  Interventions: Other: Hip flexion
- Stent (Other): Patients referred for endovascular stenting of the common femoral artery with and indication of CTA before the surgery. For these patient a CTA will be performed 1 month before and 1 month after surgery
  Interventions: Other: Hip flexion

INTERVENTIONS:
Other: Hip flexion — during the delay phase, the patients are asked to bend their knee in order to achieve the maximum degree of hip flexion

SUMMARY:
Peripheral artery diseases (PAD) are associated with an overall increased risk of mortality and morbidity, as a consequence of fatal or non-fatal vascular events, mainly due to the total or partial occlusion of the affected artery. Particularly, lower extremity occlusive arterial diseases remain a global concern, affecting more than 200 million people worldwide in 2015. Regarding the iliofemoral segment and, especially, the common femoral artery (CFA), conventional surgical approach (namely common femoral endarterectomy, CFE) is still as the gold standard despite its high morbidity rates mainly due to high rate of wound sepsis and autonomy loss . Endovascular procedures with CFA stenting have been introduced as a promising alternative for their multiple advantages such as shorter hospital stay and less perioperative complications. However, its acceptance among the vascular surgery community has been limited.

Endovascular stenting aims to reduce restenosis and improve the target lesion revascularization rates by the implementation of the stent at the level of the CFA. Nevertheless, fear of stent fracture due to hip mobility constitutes one of the main limitations to its implantation, despite the lack of widely accepted quantitative evidence of their relationship. Thus, this study aims to validate that the stresses and deformations on the iliofemoral segment during hip flexion are not a direct cause of stent fracture.

Numerical 3D models offer a non-invasive, inexpensive and personalized approach in the biomedical engineering field; thereby encouraging their use for the biomechanical study of different anatomical structures. These models are able to simulate the behavior and, additionally, quantify the forces, stresses and deformations of different organs and systems by implementing the information gathered in clinical measurements, diagnostic tests and imaging. 3D models can be reconstructed from computed tomography scans (CT scans). Specifically, CT angiography (CTA) images, offering high-quality and high-contrast images, facilitate the creation of numerical models of the vascular system (including the iliofemoral segment).

Our study will analyze the mechanical behavior of the iliofemoral segment by the creation of a numerical simulation to estimate the stresses and deformations at the level of the CFA during hip flexion. For this purpose, our project aims to use 3D models of this region reconstructed CT scans that are routinely performed preoperatively for PAD patients. Indeed CT scan are indicated for anatomical characterization of PAD lesions and guidance for optimal revascularization therapy.

The results of this study could be applied to the assessment of the treatment of lower extremities occlusive arterial diseases at the level of the CFA.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age > 65 years old
* Patient with Glomerular filtration rate > 60ml/mn
* Patient affiliated to the French Health insurance system
* Patient with a preoperative duplex scan of the lower limbs
* Patient with an indication of CT scan with either diagnostic or preoperative purposes
* Patient referred for endovascular procedure (aortic or peripheral), with an indication of CTA comprising the CFA region, without significant lesions of the external iliac and common femoral arteries (control group) or patients referred for endovascular stenting of the common femoral artery (stent group)

Exclusion Criteria:

* Patient with significant below the knee arterial lesions according the duplex scan analysis
* Hip arthroplasty.
* Hip pain and stiffness caused by hip arthritis.
* Patient under guardianship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his/her data for this research

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
deformation and stress | 6months
  a composite outcome will be used to describe both deformation and mechanical stresses from minimum to maximum hip flexion. It will comprise:
  * Variation of lumen diameter (in mm and percentage) and length of the ROI (mm).
  * Angulation (°) and maximum inscribed sphere (MIS) diameter (mm) at the bending points normalized by the degree of hip flexion as described in Figure 1A.
  * Variation of the strain (%).
  * Variation shear stresses (in mPa).
  * Variation of Von Mises stress and ,1st and 3rd principal stresses Each of these elements will be calculated at the level of the Region of Interest (ROI) measured by numerical simulation. The ROI covers the arterial segment between the section located 2cm above the inguinal ligament (end of external iliac artery) to the section located 3 cm above the crossing with the sartorius for the superficial femoral artery and 1cm above the CFA bifurcation for the deep femoral artery.

SECONDARY OUTCOMES:
anatomical variations of the artery | 6 months
  * Variation of lumen diameter (in mm and percentage) and length of the ROI (mm).
  * Angulation (°) and maximum inscribed sphere (MIS) diameter (mm) at the bending points.
Evaluation of the mechanical forces | 6months
  * Cross-sectional forces over the centerline of the ROI (Newtons) and bending moments (Newton x meter)
  * Resultant forces at contact interfaces along the ROI and boundary forces (Newtons).
Analysis of the internal and kinetic energy | 6months
  - Kinematic and internal energy (N*m) along the ROI (maximum and minimum values and localization).
Evaluation of the risk of stent fracture | 6months
  * Strain (%), shear stresses, von Mises stress and ,1st and 3rd principal stresses at the stent
  * Variation of stent's diameter (in mm and percentage) and length (mm).
  * Angulation (°) and maximum inscribed sphere (MIS) diameter (mm) at the bending points of the stent.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: No